CLINICAL TRIAL: NCT06147817
Title: Ureteroscopy With Holmium:YAG Laser Lithotripsy for Ureteral Stones in Children; What Has Changed With the Increase in Experience?
Brief Title: Ureteral Stones in Children; What Has Changed With the Increase in Experience?
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Tuğrul Tiryaki, Profesor, Director of Pediatric Urology Training, Ankara City Hospital Bilkent
Other Study IDs: E-2-23-5304
Record Dates: First submitted 2023-11-14; First posted 2023-11-28 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Ureter Stone; Childhood
Keywords: Ureter Stone; Children; Complication; Stone Free Rate
MeSH Terms: conditions — Ureterolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
With advances in endourological equipment, minimally invasive procedures have been found to be sufficient for the treatment of ureteral stones in children. The investigators aimed to evaluate the stone-free rate and complications related to the procedure and to compare it with the period when their experience were limited by presenting their patients with ureteral stones treated by ureteroscopy (URS) and holmium YAG laser in the last three years after their 15-year routine endourological practice.

The investigators retrospectively compared 54 cases treated with ureteroscopy (URS) for ureteral stones between 2009-2011, the first three years of our endourological interventions in children, and 78 cases treated with URS for ureteral stones between 2020-2022, the last three years of their 15-year endourological experience, from hospital records. Demographic data, stone-free rates, number of procedures and recorded complications were evaluated in both groups.

DETAILED DESCRIPTION:
Due to the changing diet habits and sedentary lifestyle, the investigators encountered urinary system stones more and more frequently in children. Ureteral stones in children are now routinely treated with endourological interventions with the introduction of thin ureteroscopes. Despite the developing endoscopy technology, the smaller ureter diameter in children than in adults requires more careful and meticulous intervention technically. The investigators have published that in their first 54 cases in which they started to use routine endourological methods in the treatment of ureteral stones in pediatric patients between 2009 and 2011, the investigators had a stone-free rate of 57%, a complication rate of 9.7%, and a conversion rate of 18.75% to open surgery in the first attempt. In the literature, it is seen that different results are given in terms of stone-free and complications after ureteroscopy treatment for ureteral stones in children. The investigators aimed to evaluate the stone-free rate and complications related to the procedure and compare it with the period when our experience was limited by presenting their patients with ureteral stones that the investigators treated with ureteroscopy and Holmium YAG laser in the last three years, following their 15-year-old endourological routine practice experience.

Between 01 01 2020 and 31 12 2022, 78 children with ureteral stones who were operated on in their clinic were retrospectively evaluated from the hospital records. A total of 40 males and 38 females with a mean age of 9,64+4,91 years (range 0.75 to 17) required surgical treatment for ureteral stones. USG or computerized tomography was performed in all cases, and mean stone size was 6.58+2.94 mm. (range 3,5 to 20). When stones did not pass spontaneously, the patients were treated with ureteroscopic laser lithotripsy.

All ureteroscopic procedures were performed under general anesthesia. An initial cystoscopy was done with a 8 Fr Storz cystoscope. A working guide wire was placed and negotiated beyond the level of the stone. A 4,5 Fr semirigid ureteroscope was used in all cases. Calculi were fragmented using holmium YAG laser. Fragments were extracted using a stone basket or grasper. The decision to place an ureteric stent postoperatively was based on the degree of ureteral trauma. The extracted stone fragments were sent for chemical analysis and further medical treatment initiated when appropriate. In children in whom ureteroscopy was not possible due to inability to introduce the ureteroscope, an ureteric stent was placed for passive dilation and ureteroscopy repeated 3 week later. All ureteroscopic procedures were carried out under antibiotic cover. All children underwent routine ultrasonography and urine examination in the follow-up period.

Stone-free status was determined both endoscopically at the end of the procedure and radiologically (USG) at 3 months follow-up prior to outpatient review. Stone-free rate (SFR) was defined as fragments confrmed radiologically and at least 6 months passed since the previous operation.

ELIGIBILITY:
Inclusion Criteria:

* children with ureteral stones who were operated on in our clinic

Exclusion Criteria:

* • The exclusion criteria were cases that were converted to open surgery, cases in which URS could not be performed because of anatomical reasons,

Ages: 9 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Between 01 01 2020 and 31 12 2022, 78 children with ureteral stones who were operated on in our clinic were retrospectively evaluated from the hospital records. A total of 40 males and 38 females with a mean age of 9,64+4,91 years (range 0.75 to 17) required surgical treatment for ureteral stones.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Determination of stone-free rate in children who underwent ureteroscopy (URS) for ureter stone | Ultrasonography evaluation was performed postoperative 1. month, 3-6-12-18 months, and ureter stones of the patients were evaluated.
  After the ureteroscopy, patients were monitored with Ultrasonography in the first month, 3-6-12 months, and stone-free rates were determined.
Rate of complication in children who underwent URS for ureter stone | Evaluation include postoperative 1. month
  Perioperative and postoperative complications noted
The stone-free percentages and complications percentages detected in the period when endoscopic procedures were started and in the last period when experience increased were compared. | Perioperative and postoperative first month data from two different periods will be compared
  The effect of experience on the results was determined by comparing the complications percentage and stone-free percentage of the two periods.

CONTACTS AND LOCATIONS:
Overall Officials: Huseyin T Tiryaki, MD, Study Director — University of Health Science Ankara Bilkent City Hospital
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Describe the IPD sharing plan, including what IPD are to be shared with other researchers.

REFERENCES:
- [Background] Tiryaki T, Azili MN, Ozmert S. Ureteroscopy for treatment of ureteral stones in children: factors influencing the outcome. Urology. 2013 May;81(5):1047-51. doi: 10.1016/j.urology.2013.01.008. Epub 2013 Mar 7. PMID 23465154